CLINICAL TRIAL: NCT02529150
Title: WISER After Ovarian Cancer - Exercise Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Purpose: Supportive Care
Other Study IDs: UPCC 38814
Record Dates: First submitted 2015-06-19; First posted 2015-08-20 (Estimated); Last update posted 2020-04-16 (Actual); Status verified 2020-04

CONDITIONS: Ovarian Cancer
MeSH Terms: conditions — Ovarian Neoplasms | interventions — Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- exercise (Experimental)
  Interventions: Behavioral: Exercise

INTERVENTIONS:
Behavioral: Exercise — This is an exercise intervention study. All 10 participants will complete 26 weeks high dose exercise (60% of peak aerobic capacity 45 min/session, 5 sessions per week).

SUMMARY:
One in four deaths in the United States is due to cancer, and one in three women will develop cancer in her lifetime. Despite improvements in survival among other forms of cancer, ovarian cancer prognosis remains poor. Eighty percent of women with ovarian cancer will present with advanced disease (stage 3 or 4) where 5-year survival ranges from 18-34%.2 Among patients with stage III and IV epithelial ovarian cancer (EOC), recurrence rates are high.4 Therefore, interventions focused on preventing recurrence or slowing progression of EOC is a critical problem in the field. The investigators have submitted an R21 to NCI for a dose response exercise intervention trial to examine the dose response effects of aerobic exercise on biomarkers relevant to ovarian cancer progression and recurrence. The reviewers would like assurance that the investigators can recruit ovarian cancer patients into an exercise study and that these women will do the exercise protocol we plan to prescribe in our high dose of exercise.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of stage III-IV EOC, completed surgery,
* > 12 months life expectancy (physician estimate),
* able to walk 15 minutes at a time (use of a cane is acceptable).

Exclusion Criteria:

* medical or psychiatric conditions (beyond ovarian cancer, its treatment, and its symptoms) that would impair our ability to test study hypotheses (e.g. cardiac, pulmonary, or
* orthopedic history that would prohibit a program of walking for exercise;
* psychotic disorders,
* dementia,
* inability to give informed consent

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2015-05; Primary Completion 2015-12 (Actual); Study Completion 2016-05-06 (Actual)

PRIMARY OUTCOMES:
Number of adverse events | 26 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Kathryn Schmitz, PhD, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States